CLINICAL TRIAL: NCT03387566
Title: A Phase 1, Safety, Tolerability and Pharmacokinetic Profile Study of Intravitreous Injections of HB002.1M (a Vascular Endothelial Growth Factor Receptor Decoy) in Subjects With Neovascular Age-Related Macular Degeneration
Brief Title: A Study of Single Intravitreal Injection HB002.1M in Subjects With Neovascular Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HB002.1M-01
Record Dates: First submitted 2017-12-11; First posted 2018-01-02 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Neovascular Age-Related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HB002.1M 0.3mg (Experimental): Participants received a 0.3mg dose of HB002.1M via intravitreal (IVT) injection.
  Interventions: Drug: HB002.1M
- HB002.1M 0.5mg (Experimental): Participants received a 0.5mg dose of HB002.1M via intravitreal (IVT) injection.
  Interventions: Drug: HB002.1M
- HB002.1M 1.0mg (Experimental): Participants received a 1.0mg dose of HB002.1M via intravitreal (IVT) injection.
  Interventions: Drug: HB002.1M
- HB002.1M 2.0mg (Experimental): Participants received a 2.0mg dose of HB002.1M via intravitreal (IVT) injection.
  Interventions: Drug: HB002.1M
- HB002.1M 3.0mg (Experimental): Participants received a 3.0mg dose of HB002.1M via intravitreal (IVT) injection.
  Interventions: Drug: HB002.1M

INTERVENTIONS:
Drug: HB002.1M — HB002.1M is a Vascular Endothelial Growth Factor Receptor Decoy.
  Other Names: Recombinant Human Vascular Endothelial Growth Factor Receptor-Immunoglobulin(IgG) Fc Fusion Protein Ophthalmic Injection

SUMMARY:
The objectives of this study are to evaluate the safety, tolerability, and pharmacokinetic profile of HB002.1M, a human immunoglobulin Fc fusion protein containing domain 2 and flanking sequence of vascular endothelial growth factor (VEGF) receptor-1 in subjects with age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* Age 50 to 80 years old of either gender
* Study eye must meet following requirements:

  * Active CNV lesions secondary to AMD
  * A lesion area <30 mm2 (12 disc areas) of any lesion type
  * BCVA ranging from 73-19 letters (20/32-20/400 Snellen equivalent), inclusive
  * Clear ocular media and adequate pupil dilation to permit good quality photographic imaging
* Fellow eye must have had BCVA of 19 letters ( 20/400 Snellen equivalent) or better

Exclusion Criteria:

Any ophthalmic condition as below:

* Presence of non-exudative AMD in the study eye as determined by investigator that affect macular examination, or presence of any diseases that affect central vision (including central retinal vein occlusion, diabetic retinopathy, uveitis, vascular fringes, pathological myopia, amotio retinae, macula hole etc.
* Subretinal hemorrhage in the study eye the area of hemorrhage≥of total lesion area, or hemorrhage in central fovea≥1 disc area
* Presence of scar, fibrosis or atrophy in central fovea of the study eye
* CNV of the study eye associated with other ocular conditions , such as pathologic myopia, ocular histoplasmosis, posterior uveitis, or trauma
* Anatomic damage to the center of the fovea including fibrosis and scarring making up >50% of total lesion area including the CNV in the study eye
* History or presence of a retinal pigment epithelial tear, rhegmatogenous retinal detachment or macular hole in the study eye
* History of study eye with intraocular or any ophthalmic surgery within prior 3 months (including Laser Photocoagulation at the para fovea , cataract etc.)
* History of study eye with photodynamic therapy, macular translocation surgery trabeculectomy, Recess photocoagulation, thermal laser or external beam radiation in the study eye
* History within 6 months of screening of following treatments(such as Macugen, Lucentis, Avastin, Eylea, Conbercpet, steroids etc)
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure of >25 mmHg despite treatment with maximal medical therapy)
* History of any vitreous hemorrhage within 3 months

Any systemic conditions as below:

* Currently or potentially using any drug that will cause ocular toxicity, such as psoralen, risedronic acid; or tamoxifen etc.
* Allergic to sodium fluorescein, indocyanine green, therapeutic or diagnostic protein products, and allergic to ≥ two drugs or non-drugs, or with current allergic disease
* Uncontrolled diabetes mellitus (fast glucose level ≥7.0 mmol/L or ≥11.1 mmol/L 2h after meal)
* History of surgery and/or unhealed wound, ulcer, fracture etc. 1 month prior to screening
* Any infectious disease requiring oral, intramuscular or intravenous administrations
* History of Myocardial infarction and cerebral infarction within 6 months of screening
* Active diffuse intravascular coagulation 3 months prior to screening
* Systemic immunological diseases
* Uncontrolled hypertension ≥150 mmHg systolic or ≥95 mmHg diastolic at baseline
* Any severe or uncontrolled medical conditions (eg, unstable or progressive cardiovascular, pulmonary, Parkinson, liver, or renal disease or cancer or dementia)

Any abnormal laboratory results as below:

* Abnormal liver or kidney function test value (glutamic-oxalacetic transaminase(AST), glutamic-pyruvic transaminase(ALT), creatinine(Crea), blood urea nitrogen(BUN) that was more than 1.2 times of the upper limit of normal value)
* Abnormal coagulation test(≥3 sec of upper limit value of prothrombin time, ≥10 sec of upper limit value of activated partial thromboplastin time(APTT))
* Positive in HbsAg, hepatitis C virus(HCV) antibody, human immunodeficiency virus(HIV) antibody and syphilis antibody

Other conditions related to subjects with women of childbearing potential:

* Without using any contraceptive method
* Pregnancy or lactation (urine pregnancy test positive)

Others:

* Participated clinical studies using any medications (not including vitamins and minerals) 6 months prior to screening
* Any assessment by the investigator to be unable to or unwilling to comply with requirements of the protocol

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Incidence of AE (Adverse Effect), DLT (Dose Limit Toxicity) and MTD (Maximum Tolerance Dose) | Up to 1 month after the single dose
  Incidence of AE (Adverse Effect), DLT (Dose Limit Toxicity) and MTD (Maximum Tolerance Dose)

SECONDARY OUTCOMES:
T1/2 (Terminal phase half life) after single dose | 1 months
Cmax (maximum observed concentration) after single dose | 1 months
AUC (Area Under Concentration-Time Curve) after single dose | 1 months
Immunogenicity Evaluation after single dose | 2 months
  Incidence of ADA(Anti-Drug Antibody) response
Change in Best Corrected Visual Acuity (BCVA) from baseline | 1 month
Change in central retinal thickness from baseline by Optical Coherence Tomography (OCT) | 1 month
Change in Choroidal Neovascularization (CNV) lesion area from baseline according to fluorescein angiogram | 1 month
Change of VEGF(Vascular Endothelial Growth Factor A) from baseline | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China